CLINICAL TRIAL: NCT03651011
Title: Navigated Laser In Branch Retinal Vein Occlusion Study
Acronym: NIRVANA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Danske Regioner (Other); Synoptik-Fonden (Unknown); Toyota-Fonden (Other); AP Moeller Foundation (Other); Yamagata University (Other); Queen's University, Belfast (Other); Zealand University Hospital (Other); Region Sjællands og Region Syddanmarks forskningspulje (Unknown)
Responsible Party: Principal Investigator, Katrine Hartmund Frederiksen, Principal Investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIRVANA; S-20170084 (Other: The Regional Committees on Health Research Ethics)
Record Dates: First submitted 2018-08-24; First posted 2018-08-29 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Branch Retinal Vein Occlusion; Macular Edema
Keywords: Branch Retinal Vein Occlusion; Navigated laser photocoagulation; Macular Edema; Oximetry; Retinal vascular caliber measurements; Microperimetry
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aflibercept + Navigated laser (Active Comparator): Patients will receive intravitreal aflibercept at M0, M1 and M2 (loading phase) and in addition receive navigated retinal laser photocoagulation at M3. Patients will receive aflibercept according to pro re nata regimen from M3-M12.
  Interventions: Drug: Aflibercept Injection [Eylea]; Procedure: Navigated laser photocoagulation
- Aflibercept only (Active Comparator): Patients will receive intravitreal aflibercept at M0, M1 and M2 (loading phase). Patients will receive aflibercept according to pro re nata regimen from M3-M12.
  Interventions: Drug: Aflibercept Injection [Eylea]

INTERVENTIONS:
Drug: Aflibercept Injection [Eylea] — Intravitreal injection 2 mg Eylea every 4 weeks M0-M2 (loading phase). M3-M12: continue in a pro re nata treatment regimen.
Procedure: Navigated laser photocoagulation — Navigated laser photocoagulation planned from flourscein angiography.
  Other Names: Navilas
  Arms: Aflibercept + Navigated laser

SUMMARY:
Branch retinal vein occlusion (BRVO) is often complicated by macular edema, possibly leading to severe visual loss or blindness. Treatment is repeated, intravitreal injections of vascular endothelial growth factor (VEGF)-inhibitors like aflibercept. The treatment is effective, but a need for repetitive injections is a concern for patients as well as society due to risk of side effects, regular hospital visits and the price of the drug. Former treatment included macular grid pattern photocoagulation, but this technology was limited by a poorer visual outcome for the patient and a higher risk of side effects, including central visual loss.

A novel laser delivery system, called navigated laser photocoagulation, has proven effective, safe and precise, and has shown promising results in stabilising the effect of the VEGF-inhibitor treatment in similar diseases.

Thus, in a 12-month prospective, randomized 1:1 study of 60 patients with BRVO and macular edema the investigators aim to (1) Examine the treatment response of patients treated with intravitreal aflibercept (Eylea®) and navigated retinal laser (Navilas®)(Group 1) as compared to patients treated with intravitreal aflibercept only (Group 2), and (2) Identify non-invasive retinal biomarkers (retinal oxygen saturation, macular ischemia and retinal vascular arteriolar and venular calibre) for successful treatment outcome.

DETAILED DESCRIPTION:
Purpose of the study

In a 12-month prospective, randomized 1:1 study of patients with branch retinal vein occlusion (BRVO) and macular edema, the investigators aim to

1. Examine the treatment response of patients treated with intravitreal aflibercept (Eylea®) and navigated retinal laser (Navilas®)(Group 1) as compared to patients treated with intravitreal aflibercept only (Group 2), and
2. Identify non-invasive retinal biomarkers (retinal oxygen saturation, macular ischemia and retinal vascular arteriolar and venular calibre) for successful treatment outcome.

Problem statement

Severe visual loss or blindness in BRVO is often caused by macular edema. Until a few years ago, treatment included observation or macular grid pattern laser photocoagulation. With this treatment it was often possible to stabilize the disease in a few treatment sessions. However, in recent years better visual outcome has been demonstrated with intravitreal injections of vascular endothelial growth factor (VEGF) inhibitors like ranibizumab or aflibercept. Even though this is encouraging, patients on average need nine injections in the first 12 months. The high number of repetitive treatments is a concern for patients as well as society due to the invasiveness of the treatment and the price of the drug. Hence, it is warranted to develop newer treatment regimens combining the efficacy of intravitreal anti-VEGF with the potential stabilizing effect of macular laser photocoagulation. This would be an approach that might minimize the number of injections and its side effects while still providing acceptable visual outcomes for the patients.

In addition to providing the optimal treatment, it is important to identify non-invasive markers of disease activity and treatment outcome in order to enable individualised and personalised treatment while providing novel research opportunity in this potentially blinding disease.

Theoretical foundation (Literature background)

Retinal vein occlusion (RVO) is a common cause of visual loss in the elderly with a 15-year incidence of 2.3% of the population. The condition is classified anatomically according to the site of the occlusion. Seventy eight percent of patients have an occlusion of a branch vein, which is often complicated by macular edema, leading to visual impairment.

Branch retinal vein occlusion is diagnosed based on intraretinal hemorrhages in the retinal sector drained by the affected vein. In time, hemorrhages often resorb, but vision-threatening complications may arise. The common link for these is ischemia, that leads to an upregulation of VEGF, which then causes neovascularization, vasodilation and increased vascular permeability, leading to macular edema, the most common reason for vision loss in BRVO.

With ischemia in mind, measurements of retinal oxygen saturation could provide important information regarding the metabolic status of the inner retina. The vascular oxygen saturation of the inner retina is a functional marker, that can be measured non-invasively by a spectrophotometric retinal oximeter. Even though this has only been studied on a very limited basis in BRVO, proof-of-concept has been established by Lin et al. and Hardarson et al., demonstrating cross-sectional changes in retinal oxygen saturation. However, they did not correlate these to treatment outcome.

Ischemia can also be evaluated as a structural marker. The most reliable way of evaluating this is to measure the area of retinal non-perfusion by fundus fluorescein angiography. Non-perfusion has been demonstrated as a strong marker of disease severity, but it is still uncertain if this is reversible, and if so, if this surrogate marker of VEGF-activity can potentially be used to guide the treatment.

Retinal vascular calibre is another non-invasive method of evaluating the retinal vascular system. The research unit have performed validated, semiautomatic measurements of the retinal arteriolar and venular diameters in studies of diabetic retinopathy, and demonstrated cross-sectional associations as well as longitudinal predictions of intra- and extraocular microvascular complications of type 1 diabetes. For instance, Broe et al. demonstrated that patients with narrower arterioles and wider venules had an independently higher risk of developing various microvascular complications in a 16-year prospective study. This emphasizes the importance of structural retinal changes in relation to the metabolic function. In BRVO, Youm et al. demonstrated that patients with BRVO had narrowing of retinal arterioles and venules, but any potential correlation to treatment outcome has not been examined.

Current state of the art In 1984 the Branch Vein Occlusion Study for macular edema demonstrated that 63% of patients treated with macular laser gained two or more lines of vision, compared to 36% of untreated eyes. Based on this, the standard treatment for many years was to perform macular laser photocoagulation if vision had not improved after 3-6 month of observation. However, the introduction of VEGF-inhibitors within the last decade has changed the landscape dramatically. Randomized, controlled studies like BRAVO and VIBRANT demonstrated a higher efficacy of ranibizumab and aflibercept versus sham and laser with 53-61% of patients gaining at least three lines of vision.

In Denmark, the present guidelines for treatment of BRVO with macular edema has been set in September 2015 by "Rådet for Anvendelse af Dyr Sygehusmedicin". The council recommended that intravitreal aflibercept or ranibizumab should be used as first line of treatment. However, the council also raised concern, stating that they expected an annual increment of approximately 600 new patients with RVO in Denmark putting both financial and societal burden on the individual and the healthcare system. With the chronic nature of the disease in mind, this is expected to put a significant weight on the healthcare system for the years to come.

Choice of methods

Navigated laser photocoagulation is the cornerstone of the present study. This is a novel laser delivery system that holds many advantages as compared to traditional macular laser photocoagulation. Navigated laser makes treatment easier to plan, perform and document.

Firstly, it includes an eye tracking system, which makes it safe to treat close to the foveal center. For a traditional laser it is recommended to keep a minimum distance of 500μm from the foveal center in order to limit the risk of severe visual loss. For safety reasons many physicians prefer to keep an even larger distance, which often limits the beneficial effect of the treatment. Secondly, the navigated laser system is automatic which improves the accuracy to target focal lesions by 27%. Thirdly, navigated laser makes it possible to import images from fluorescein angiographys and allows for clear delineation and consequent treatment of the diseased microvasculature.

Hypothesis

The investigators hypothesize that:

1. As compared to intravitreal aflibercept monotherapy, combination treatment with intravitreal aflibercept and navigated laser leads to a lesser number of intravitreal injections needed to stabilise vision in patients with BRVO and macular edema.
2. It is possible to use non-invasive retinal markers to predict disease activity and treatment outcome in patients with BRVO and macular edema. Regardless of treatment regimen, the investigators believe that patients who respond well to treatment will have (1) lower retinal venular oxygen saturation, (2) less macular ischemia, and (3) lower retinal venular calibre.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BRVO with foveal center-involved macular edema in the study eye.
* Best-corrected visual acuity (BCVA) 35-80 Early Treatment Diabetic Retinopathy Study (ETDRS) letters (0.1-0.8 Snellen equivalent) in the study eye at baseline (BL).
* Age ≥18 years.
* Central retinal thickness > 300 μm in the study eye at BL.
* Onset ≤ 6 months prior to the study.

Exclusion Criteria:

* Active retinal or iris neovascularizations in the study eye at any time.
* Cataract, vitreous hemorrhage or other clouding conditions that prevent retinal laser photocoagulation in the study eye at M3.
* Prior anti-VEGF treatment or macular laser photocoagulation in the study eye.
* Macular edema and/or increased retinal thickness due to other potential causes than BRVO
* Uncontrolled hypertension (blood pressure ≥ 160/110 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Patients with additional need for anti-VEGF after loading phase | Month 3 to Month 12
  Percentage of patients in Groups 1 and 2 that receive additional intravitreal aflibercept after the loading phase

SECONDARY OUTCOMES:
Additional need for anti-VEGF after loading phase | Month 3 to Month 12
  Median number of additional intravitreal aflibercept after the loading phase
Change in BCVA according to treatment regimen | Month 12
  Median change in best-corrected visual acuity (BCVA) from baseline (BL) to month (M) 12 in Group 1 and 2.
Effect on macular edema according til treatment regimen | Month 12
  Ratio of patients without macular edema at M12 in Groups 1 and 2
Retinal oxygen saturation | Baseline
  Evaluation of retinal oxygen saturation at BL as marker of disease activity and successful treatment outcome (as defined by no need for intravitreal aflibercept at M11 and M12)
Macular ischemia (area of FAZ) | Baseline
  Evaluation of macular ischemia (as determined by area of the Foveal Avascular Zone (FAZ)) at BL as a marker of disease activity and successful treatment outcome (as defined by no need for intravitreal aflibercept at M11 and M12)
Vessel geometry | Baseline
  Evaluation of retinal venular calibre at BL as a marker of disease activity and successful treatment outcome (as defined by no need for intravitreal aflibercept at M11 and M12)
Visual field | Baseline and Month 12
  Change in central visual fields, as evaluated by microperimetry according to treatment regimen

CONTACTS AND LOCATIONS:
Overall Officials: Katrine H Frederiksen, PhD-student, Principal Investigator — Research Unit of Ophthalmology, University of Southern Denmark; Jakob Grauslund, DMSci,PhD, Study Director — Research Unit of Ophthalmology, University of Southern Denmark; Torben L Sørensen, DMSci, Study Chair — Dept. of Ophthalmology, Zealand University Hospital; Jesper P Vestergaard, MD, Study Chair — Dept. of Ophthalmology, Odense University Hospital; Inger C Munch, PhD, Study Chair — Dept. of Ophthalmology, Zealand University Hospital; Tunde Peto, PhD, Study Chair — Queen's University, Belfast, England; Ryo Kawasaki, PhD, Study Chair — Yamagata, University, Japan
Locations (2):
- Denmark (2):
  - Department of Ophthalmology, Odense University Hospital, Odense, Danmark
  - Department of Ophthalmology, Zealand University Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Argon laser scatter photocoagulation for prevention of neovascularization and vitreous hemorrhage in branch vein occlusion. A randomized clinical trial. Branch Vein Occlusion Study Group. Arch Ophthalmol. 1986 Jan;104(1):34-41. doi: 10.1001/archopht.1986.01050130044017. PMID 2417579
- [Background] Brown DM, Campochiaro PA, Bhisitkul RB, Ho AC, Gray S, Saroj N, Adamis AP, Rubio RG, Murahashi WY. Sustained benefits from ranibizumab for macular edema following branch retinal vein occlusion: 12-month outcomes of a phase III study. Ophthalmology. 2011 Aug;118(8):1594-602. doi: 10.1016/j.ophtha.2011.02.022. PMID 21684606
- [Background] Pielen A, Mirshahi A, Feltgen N, Lorenz K, Korb C, Junker B, Schaefer C, Zwiener I, Hattenbach LO; RABAMES Study Group. Ranibizumab for Branch Retinal Vein Occlusion Associated Macular Edema Study (RABAMES): six-month results of a prospective randomized clinical trial. Acta Ophthalmol. 2015 Feb;93(1):e29-37. doi: 10.1111/aos.12488. Epub 2014 Jul 8. PMID 25042729
- [Background] Clark WL, Boyer DS, Heier JS, Brown DM, Haller JA, Vitti R, Kazmi H, Berliner AJ, Erickson K, Chu KW, Soo Y, Cheng Y, Campochiaro PA. Intravitreal Aflibercept for Macular Edema Following Branch Retinal Vein Occlusion: 52-Week Results of the VIBRANT Study. Ophthalmology. 2016 Feb;123(2):330-336. doi: 10.1016/j.ophtha.2015.09.035. Epub 2015 Oct 30. PMID 26522708
- [Background] Klein R, Moss SE, Meuer SM, Klein BE. The 15-year cumulative incidence of retinal vein occlusion: the Beaver Dam Eye Study. Arch Ophthalmol. 2008 Apr;126(4):513-8. doi: 10.1001/archopht.126.4.513. PMID 18413521
- [Background] Aiello LP, Avery RL, Arrigg PG, Keyt BA, Jampel HD, Shah ST, Pasquale LR, Thieme H, Iwamoto MA, Park JE, et al. Vascular endothelial growth factor in ocular fluid of patients with diabetic retinopathy and other retinal disorders. N Engl J Med. 1994 Dec 1;331(22):1480-7. doi: 10.1056/NEJM199412013312203. PMID 7526212
- [Background] Noma H, Minamoto A, Funatsu H, Tsukamoto H, Nakano K, Yamashita H, Mishima HK. Intravitreal levels of vascular endothelial growth factor and interleukin-6 are correlated with macular edema in branch retinal vein occlusion. Graefes Arch Clin Exp Ophthalmol. 2006 Mar;244(3):309-15. doi: 10.1007/s00417-004-1087-4. Epub 2005 Aug 13. PMID 16133018
- [Background] Geirsdottir A, Palsson O, Hardarson SH, Olafsdottir OB, Kristjansdottir JV, Stefansson E. Retinal vessel oxygen saturation in healthy individuals. Invest Ophthalmol Vis Sci. 2012 Aug 13;53(9):5433-42. doi: 10.1167/iovs.12-9912. PMID 22786895
- [Background] Lin LL, Dong YM, Zong Y, Zheng QS, Fu Y, Yuan YG, Huang X, Qian G, Gao QY. Study of retinal vessel oxygen saturation in ischemic and non-ischemic branch retinal vein occlusion. Int J Ophthalmol. 2016 Feb 18;9(1):99-107. doi: 10.18240/ijo.2016.01.17. eCollection 2016. PMID 26949618
- [Background] Hardarson SH, Stefansson E. Oxygen saturation in branch retinal vein occlusion. Acta Ophthalmol. 2012 Aug;90(5):466-70. doi: 10.1111/j.1755-3768.2011.02109.x. Epub 2011 Apr 21. PMID 21518303
- [Background] Grauslund J, Hodgson L, Kawasaki R, Green A, Sjolie AK, Wong TY. Retinal vessel calibre and micro- and macrovascular complications in type 1 diabetes. Diabetologia. 2009 Oct;52(10):2213-7. doi: 10.1007/s00125-009-1459-8. Epub 2009 Jul 18. PMID 19618163
- [Background] Broe R, Rasmussen ML, Frydkjaer-Olsen U, Olsen BS, Mortensen HB, Hodgson L, Wong TY, Peto T, Grauslund J. Retinal vessel calibers predict long-term microvascular complications in type 1 diabetes: the Danish Cohort of Pediatric Diabetes 1987 (DCPD1987). Diabetes. 2014 Nov;63(11):3906-14. doi: 10.2337/db14-0227. Epub 2014 Jun 9. PMID 24914239
- [Background] Youm DJ, Ha MM, Chang Y, Song SJ. Retinal vessel caliber and risk factors for branch retinal vein occlusion. Curr Eye Res. 2012 Apr;37(4):334-8. doi: 10.3109/02713683.2011.629070. Epub 2012 Feb 10. PMID 22324736
- [Background] Techniques for scatter and local photocoagulation treatment of diabetic retinopathy: Early Treatment Diabetic Retinopathy Study Report no. 3. The Early Treatment Diabetic Retinopathy Study Research Group. Int Ophthalmol Clin. 1987 Winter;27(4):254-64. doi: 10.1097/00004397-198702740-00005. No abstract available. PMID 3692707
- [Background] Kozak I, Oster SF, Cortes MA, Dowell D, Hartmann K, Kim JS, Freeman WR. Clinical evaluation and treatment accuracy in diabetic macular edema using navigated laser photocoagulator NAVILAS. Ophthalmology. 2011 Jun;118(6):1119-24. doi: 10.1016/j.ophtha.2010.10.007. Epub 2011 Jan 26. PMID 21269701
- [Background] Tomkins-Netzer O, Ismetova F, Bar A, Seguin-Greenstein S, Kramer M, Lightman S. Functional outcome of macular edema in different retinal disorders. Prog Retin Eye Res. 2015 Sep;48:119-36. doi: 10.1016/j.preteyeres.2015.05.002. Epub 2015 May 23. PMID 26014685
- [Background] Liegl R, Langer J, Seidensticker F, Reznicek L, Haritoglou C, Ulbig MW, Neubauer AS, Kampik A, Kernt M. Comparative evaluation of combined navigated laser photocoagulation and intravitreal ranibizumab in the treatment of diabetic macular edema. PLoS One. 2014 Dec 26;9(12):e113981. doi: 10.1371/journal.pone.0113981. eCollection 2014. PMID 25541960
- [Derived] Frederiksen KH, Pedersen FN, Vergmann AS, Yang D, Laugesen CS, Vestergaard JP, Sorensen TL, Cheung CY, Kawasaki R, Peto T, Grauslund J. Predictive value of retinal oximetry, optical coherence tomography angiography and microperimetry in patients with treatment-naive branch retinal vein occlusion. Int J Retina Vitreous. 2023 Jun 28;9(1):38. doi: 10.1186/s40942-023-00468-7. PMID 37381014